CLINICAL TRIAL: NCT01539369
Title: A Study to Investigate the Short and Long Term Effects of Two 12-week Healthy Eating Interventions on Body Weight, Body Composition, Appetite Control, Biomarkers of Health and Subjective Wellbeing in Overweight Women
Brief Title: The Leeds Women's Wellbeing (LWW) Study
Acronym: LWW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Prof Louise Dye, Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 10/H1305/6
Record Dates: First submitted 2011-12-02; First posted 2012-02-27 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Weight Loss
Keywords: dietary intervention; dietary fibre; weight loss; weight maintenance
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fibre diet (Experimental)
  Interventions: Other: Healthy eating diet (Diet A) or healthy eating diet combined with advice to increase fibre intake (Diet B) to at least 25g/day
- Healthy eating diet (Active Comparator)
  Interventions: Other: Healthy eating diet (Diet A) or healthy eating diet combined with advice to increase fibre intake (Diet B) to at least 25g/day

INTERVENTIONS:
Other: Healthy eating diet (Diet A) or healthy eating diet combined with advice to increase fibre intake (Diet B) to at least 25g/day — Participants were randomly assigned to one of two parallel arms:
  Diet A:healthy eating without extra advice to increase fibre intake or Diet B: healthy eating with extra advice to increase fibre intake to a minimum of 25g/d. Healthy eating advice was based on the British Heart Foundation booklet: "Food Should Be Fun And Healthy". Participants following Diet A were encouraged to eat breakfast cereals and were provided with complementary cereals and snacks low in fibre. Participants following Diet B were encouraged to eat high fibre breakfast cereals and to incorporate wheat bran fibre in other meals. Complementary high fibre cereals and snacks were provided.

SUMMARY:
The purpose of this parallel design study is to assess the relative effects of two 12-week healthy eating dietary interventions: general healthy eating (Diet A) and general healthy eating combined with advice to increase fibre intake (Diet B) to at least 25g/day (with a large proportion of the fibre intake derived from cereal or wheat bran), in overweight low-fibre consuming premenopausal female adults on body weight change (kg). It is hypothesized that adding fibre to a healthy eating diet (Diet B) would lead to greater weight loss and/or weight loss maintenance than following a healthy eating diet alone (Diet A).

DETAILED DESCRIPTION:
In this randomised, single blind, parallel design study participants were randomly assigned to one of two 12-week healthy eating dietary interventions: Diet A: general healthy eating OR Diet B: general healthy eating combined with advice to increase fibre intake to at least 25g/day (with a large proportion of the fibre intake derived from cereal or wheat bran.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-48 years of age (premenopausal)
* Self reported good health
* Body Mass Index (BMI) within overweight/obese range (26-35kg/m2)
* Willingness to consume study foods and prepared to eat breakfast cereals as part of the intervention
* Non-smokers or given up more than 6 months ago
* Exercising no more than 4 times per week at a medium intensity
* Weight stable in the last 3 months (fluctuation of no more than 3kg)
* Current fibre intake (≤ 15g/day) according to DINE and verified by 7 day food diary (fibre points)
* Ability to adequately understand verbal and written information in English

Exclusion Criteria:

* Menopausal or showing menopausal symptoms (e.g. frequent/recurrent hot flushes) at screening or taking any supplements for menopausal symptoms
* Type 2 Diabetes; Cardiac pacemaker fitted
* Taking medication and/or supplements known to affect appetite/body weight in the last 6 months (e.g. asthma, steroids, anti-depressants)
* BMI outside range of 26-35 kg/m2
* Food allergies or aversions to foods likely to be consumed within the study (e.g. wheat bran, nuts)
* Non-smokers or given up more than 6 months ago
* Exercising more than 4 times per week at a medium intensity
* Shift work (night shifts)
* Pregnant or planning a pregnancy within the next year; having been pregnant or lactating within the previous 6 months
* No history of, or current eating disorders as determined using the Eating Attitudes Test (EAT-26;Gardner et al., 1982; a score higher than 20)
* Current fibre intake (>15g/day according to DINE)
* Insufficient English language skills to complete all study questionnaires

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
body weight change (kg) during the 12 week intervention | at screening and every 4 weeks at each subsequent visit, the last week of the intervention (week 12), at one month and one year after the intervention has finished
  Body weight will be measured three times using ADP (BodPod, Concord, CA, USA); once during the inclusion phase (week -1), at the end of the intervention (week 12) and at follow up (one year later). Body weight will also be measured six times using bioimpedance (Tanita, Illinois, USA); once during the inclusion phase (week -1) and then again during weeks 4, 8, 12 of the intervention phase and at follow up (one month later and one year later)

SECONDARY OUTCOMES:
Food Intake | 7 day food diary the week before starting the intervention; 3 day food diaries at baseline (first week of the intervention), then baseline +4 weeks, baseline +8 weeks, baseline +12 weeks, baseline +12 months
  A 7-day food intake diary (self-reported food intake using household measures) will be completed during the first week of the inclusion phase to allow an assessment of habitual daily energy, macronutrient and fibre intake. Three-day food intake diaries (self-reported food intake using household measures on 2 weekdays and 1 weekend day) will be completed during study weeks 1, 5, 9, 12 and at one year follow up
Glycaemic regulation | at baseline (first week of the intervention over a period of 3 days) and at baseline +12 weeks (last week of the intervention over a period of 3 days)
  This will be assessed using continuous glucose monitoring (CGMS) in a subsample of participants N=24, with N=12 from each treatment arm. Fasting measures of insulin and glucose will be obtained to assess Homeostasis Model Assessment (HOMA) and diabetes risk before and at the end of the intervention
Biochemical measures | at baseline (first week of the intervention) and then at baseline +12 weeks (last week of the intervention)
  Fasting blood samples will be collected during the first week of the intervention and in the last week of the intervention (week 12) on the morning of a test meal challenge day. These fasting samples will be assayed for glucose, insulin, cholesterol, triglycerides and also leptin. These blood samples will be collected at the phlebotomy outpatient clinic at the Leeds General Infirmary. Further blood samples, which will be assayed for appetite hormones (Ghrelin, GLP-1, PYY and CCK), will be taken pre and post lunch on the test meal challenge days via a cannula fitted by a research nurse.
Subjective symptoms, wellbeing and Mood | Wellbeing Diary Booklets (WDBs) will be completed each day from screening till the last week of the intervention (week 12)
  Each day women will complete a symptom checklist which will ask them to rate a range of symptoms on a five point Likert Scale from 0 (none) to 4 (extreme). The checklist will comprise items relating to women's general wellbeing (e.g. digestive sensations, mood and wellbeing). Women will note down whether they are menstruating. Participants on Diet B will record the amount of fibre they have consumed using a points-based system, as a measure of compliance. Each day all women will be asked to complete the Bristol Stool Form Scale (BSFQ; O'Donnell et al., 1990)
Sleep and body shape perception | at baseline (first week of the intervention), baseline +4 weeks, baseline +8 weeks, baseline +12 weeks, baseline +16 weeks and then at baseline +12 months
  Participants will be asked to complete an adapted version of the Leeds Sleep Evaluation Questionnaire (LSEQ; Parrott and Hindmarch, 1978) and Body Shape Questionnaire (BSQ-34; Cooper et al, 1987) during the visits at weeks -1, 4, 12 and at one month and at one year follow up
Eating behaviour | at baseline (first week of the intervention), baseline +4 weeks, baseline +8 weeks, baseline +12 weeks, baseline +16 weeks and then at baseline +12 months
  Eating behaviour will be assessed using the Dutch Eating Behaviour Questionnaire (DEBQ; van Strien et al., 1986) and the Three Factor Eating Questionnaire (TFEQ; Stunkard and Messick, 1985) at weeks 1, 4 , 8, 12 and at follow up (one month and one year later) to provide measures of dietary restraint and other psychological aspects of eating behaviour. At follow up (one year later) participants will also be asked to complete the Intuitive Eating Scale (IES; Tylka, 2006) in order to measure the levels of intuitive eating behaviour
Diet Satisfaction | at baseline +12 months
  The Diet Satisfaction questionnaire (D-SAT; Ello-Martin et al., 2004) to assess participants satisfaction with their current diet
Depression Anxiety and Stress | at baseline +12 months
  The Depression Anxiety Stress Scale (DAAS42; Lovibond and Lovibond,1995) will be used to assess depression anxiety and stress at one year follow up in order to assess symptoms of depression, anxiety and stress.
Life events | at baseline +12 months
  Participants will be asked to complete the Social Readjustment Rating Scale (SRRS) also known as Life Events Scale (LES; Holmes and Rahe, 1967) in order to assess stressful events that they may have experienced over the last 12 months
Dietary fibre intake | at recruitment visit, at baseline +12 weeks, at baseline +16 weeks and at baseline +12 months
  Participants will be asked to complete the Dietary Instrument for Nutrition Education (DINE; Roe et al., 1994) and the Leeds Women's Wellbeing Fibre Intake Assessment (LWW-FIA) to assess habitual fibre intake catergorically (DINE) and in grams/day (LWW-FIA)
body composition | at baseline (first week of the intervention), baseline +4 weeks, baseline +8 weeks, baseline +12 weeks, baseline +16 weeks and then at baseline +12 months
  Body composition will be measured four times using ADP (BodPod, Concord, CA, USA), once during the inclusion phase (week -1), once during the last week of the intervention (week 12) and at follow up (one month and one year later). Body composition will also be measured six times using bioimpedance (Tanita, Illinois, USA) at the inclusion phase (week -1), at weeks 4, 8, 12 of the intervention and at follow up (one month later and one year later).
Waist circumference | at baseline (first week of the intervention), baseline +4 weeks, baseline +8 weeks, baseline +12 weeks, baseline +16 weeks and then at baseline +12 months
  Waist circumference will be taken six times according to established methods (Van der Kooy and Seidell, 1993) during the inclusion phase (week -1), at weeks 4,8,12 of the intervention and at follow up (one month later and one year later).
Appetite ratings | Five times over a period of 2 hours during a test meal challenge day once at the beiginning of the intervention (baseline) and once at the end of the intervention (baseline +12 months)
  100mm Visual Analogue Scale (VAS) ratings of subjective motivation to eat (hunger, fullness, desire to eat and prospective consumption) were completed before and 4 times after a fixed energy lunch meal during the first week of the intervention and then again at the end of the intervention
Food preferences | Before and after consumption of a fixed energy test meal at baseline (first week of the intervention) and again before and after the second test meal at the last week of the intervention (baseline + 12 months)
  The Food Preference Checklist (FPC; Blundell and Rogers, 1980) will be completed before and immediately after consumption of the fixed energy test meal

CONTACTS AND LOCATIONS:
Overall Officials: Louise Dye, Professor, Principal Investigator — University of Leeds
Locations (1):
- Institute of Psychological Sciences, Leeds, United Kingdom